CLINICAL TRIAL: NCT05987917
Title: Clinical and Histological Evaluation of BTL-785F Non-invasive Treatment for Facial Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS300
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-08

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Group RF+USN (Experimental): Subjects will be enrolled for an active treatment with BTL-785F (BTL-785-2 applicator) delivering radiofrequency (RF) and ultrasound (USN) for non-invasive facial rejuvenation
  Interventions: Device: BTL-785-2
- Group RF (Experimental): Subjects will be enrolled for an active treatment with BTL-785F (BTL-785-2 applicator) delivering radiofrequency (RF) only for non-invasive facial rejuvenation
  Interventions: Device: BTL-785-2
- Control (Experimental): Control subject will not receive treatment
  Interventions: Other: No Treatment

INTERVENTIONS:
Device: BTL-785-2 — Treatment with BTL-785 device (BTL-785-2 applicator) for non-invasive facial rejuvenation
  Arms: Group RF; Group RF+USN
Other: No Treatment — The subject who will serve as control will not be treated with the study device.
  Arms: Control

SUMMARY:
This study will evaluate the clinical efficacy, safety and the performance of the BTL-785-2 applicator of the BTL-785F system for non-invasive treatment of facial wrinkles and correcting facial skin laxity.

DETAILED DESCRIPTION:
The changes in the skin tissue related to the levels of hyaluronic acid (HA) will be assessed histologically. The study is a prospective, single-center, three-arm, open-label study. The subjects will be enrolled and assigned into two treatment groups; group A (RF & USN) and B (only RF) which will receive a treatment with different settings. Subjects of both groups will be required to complete four (4) treatment visits and two follow-up visits. Additionally, a Control will be included to verify the treatment outcomes.

At the baseline visit, health status will be assessed. Inclusion and exclusion criteria will be verified and informed consent will be signed. Punch biopsies of the facial skin for the examination of changes related to HA levels and photographs of the treated area will be taken.

The treatment administration phase in both treatment groups will consist of four (4) treatment visits, delivered 7 - 14 days apart.

ELIGIBILITY:
Inclusion criteria

* Healthy male or female subjects over 21 years of age seeking treatment with non-invasive radiofrequency and ultrasound treatment for facial rejuvenation
* Subjects should be able to understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible wrinkles in the treated area when the face is relaxed as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits and to undergo punch biopsies in the infraauricular area.
* Agreement to have their photographs taken for the purpose of this clinical investigation.

Exclusion criteria

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Sensitivity disorders in the treatment area
* Varicose veins, pronounced edemas
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use anti-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study
* Any disease or condition contradicting the skin tissue biopsy
* Any disease or condition that may compromise the histologic observation at the pathologist discretion

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Histological examination | 5 months
  Evaluation of the facial skin tissue to assess the changes related to levels of HA in the biopsies obtained from both treatment groups and control.

SECONDARY OUTCOMES:
Subject Satisfaction | 5 months
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for evaluating the satisfaction. The Subject Satisfaction Questionnaire will be given to subjects after the last therapy, at 1-month and 3-month follow-up. The answers to the questions related to the subjects' overall skin and face appearance will vary from "strongly agree" to "strongly disagree".
Therapy Comfort | 5 months
  The 5-point Likert scale Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. Pain sensation will be rated by the subjects from 0 (no pain) to 10 (worst possible pain).
Evaluation of Wrinkle Severity | 5 months
  Three independent evaluators will evaluate changes of wrinkle severity according to the Fitzpatrick Wrinkle and Elastosis Scale (FWES) using the photographs of treated areas for wrinkles (left and right cheeks and the forehead) taken at the baseline, last therapy visit and each follow-up visit. Wrinkle severity improvement according to FWES is considered when there is a decrease in score of the scale. The baseline and post-treatment scores will be compared. If applicable, the statistical significance of obtained results will be analyzed in Microsoft Excel spreadsheet software. The level of significance (α) will be set as 5%.
Evaluation of Overall Facial Appearance According to GAIS | 5 months
  Three evaluators will evaluate facial appearance in the treatment group according to the Global Aesthetic Improvement Scale (GAIS) using the photographs taken at the baseline, last therapy visit and both follow-up visits. Each evaluator will be asked to assign a score to a set of photographs. Facial appearance improvement to GAIS is considered when there is an increase in score of the scale. The baseline and post-treatment scores will be compared. If applicable, the statistical significance of obtained results will be analyzed in Microsoft Excel spreadsheet software. The level of significance (α) will be set as 5%.

CONTACTS AND LOCATIONS:
Locations (1):
- Schweiger Dermatology PC, Reseach Division, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg DJ. A Novel Technology to Boost Natural Production of Hyaluronic Acid in the Skin Tissue: Human Histology Study. J Cosmet Dermatol. 2025 Apr;24(4):e70159. doi: 10.1111/jocd.70159. PMID 40243133